CLINICAL TRIAL: NCT03365375
Title: Mindfulness-Based Stress Reduction for Adults With Low-Risk Chest Pain Associated With Anxiety: A Pilot Trial
Brief Title: Mindfulness-Based Stress Reduction for Adults With Low-Risk Chest Pain Associated With Anxiety
Acronym: MBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Paul Musey, Assistant Professor of Emergency Medicine, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VFR-447 Musey
Record Dates: First submitted 2017-11-27; First posted 2017-12-07 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-05

CONDITIONS: Chest Pain; Anxiety; Mindfulness
Keywords: Chest Pain; Anxiety; Mindfulness; Emergency Service, Hospital
MeSH Terms: conditions — Chest Pain; Anxiety Disorders; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Referral (Active Comparator): Subjects will be referred for primary care provider (PCP) follow up and/or to psychiatry for further management and treatment of elevated anxiety levels according to standard of care.
  Interventions: Other: Usual Care Referral
- MBSR Referral (Experimental): Referral to a local mindfulness-based stress reduction course in addition to referral to their PCP.
  Interventions: Behavioral: MBSR Referral; Other: Usual Care Referral

INTERVENTIONS:
Behavioral: MBSR Referral — Referral for mindfulness-based stress reduction (MBSR), a structured meditation training program consisting of 8 weekly group sessions.
  Other Names: MBSR
  Arms: MBSR Referral
Other: Usual Care Referral — Referral to PCP or Psychiatry

SUMMARY:
This Emergency Department based study investigates the feasibility and effectiveness of a mindfulness based stress reduction (MBSR) training program referral for patients with chest pain at low risk for acute coronary syndrome but associated with anxiety. Outcomes assessed for eligible patients randomized to MBSR vs. usual care include mental health (longitudinal Generalized Anxiety Disorder - 7 (GAD-7) scores), quality of life (PROMIS Global Short Form), and ED resource utilization (return Emergency Department (ED) visits).

DETAILED DESCRIPTION:
To determine the effect of an MBSR training program for patients with low-risk chest pain associated with anxiety on mental health (longitudinal GAD-7 scores, quality of life (PROMIS Global Short Form), and ED resource utilization (return ED visits). The working hypothesis is that early referral to MBSR will help patients better regulate their thoughts, feelings, and bodily sensations related to their anxiety symptoms and have a significant positive effect on patient-centered outcomes such as mental health, quality of life as well as decreased ED resource utilization. To this end the investigators will randomize patients identified via a two step process (HEART Score <4 and GAD-7 score > 9 to usual care referrals versus MBSR. The investigators will then follow these participants for outcomes including change in GAD-7 scores, PROMIS Global Short Form, ED utilization among other outcomes at 6 weeks, 3 months, 6 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of chest pain
* HEART Score of 0-3 indicating Major Adverse Cardiac Events (MACE) risk equivalent to ≤2%
* GAD-7 score > or = 10

Exclusion Criteria:

* Age <18 or ≥ 71
* Chief complaint of anxiety, panic, or similar
* Prior personal acute coronary syndrome (ACS) history (known at time of provider interview)
* Previous enrollment in the study
* Traumatic injury to the chest
* Suicidal ideation or active psychosis or behavioral issues requiring psychiatric monitoring
* Hemodynamic instability
* Non-English speaking
* Potential issues affecting follow up: Prisoners, homeless patients, out-of-town residences

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul I Musey, MD, MS, Principal Investigator — Indiana University School of Medicine, Department of Emergency Medicine
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from the clinical study report and the study protocol will be shared upon request.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available for 5 years after study completion date.
Access Criteria: email PI at pmusey@iu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We screened patients who presented to the Emergency Department (ED) with chest pain. We assessed their risk for major adverse cardiac events (MACE) using the HEART score and for anxiety with the GAD-7. Enrolled subjects were assigned to either arm depending upon enrollment period. In the 8 weeks prior to the MBSR course commencement all subjects enrolled were assigned to Arm 2: MBSR. This period was immediately followed by 8 weeks of enrollment in Arm 1: Standard Referral.
Period: Overall Study
Arm/Group | Usual Care Referral | MBSR Referral
Started | 14 | 14
Completed | 14 | 9
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Referral | MBSR Referral | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (9.3) | 38.9 (11.9) | 41.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
GAD-7 at enrollment [Mean (Standard Deviation); unit: units on a scale] | 15.9 (4.4) | 14.9 (3.1) | 15.3 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Generalized Anxiety Disorder -7 (GAD-7)
Description: Difference in GAD-7 score at enrollment compared to assessment at 3 months. Anxiety Severity by total score. Range 0-21. Mild 5-9; Moderate (10-14); Severe > 15
Time Frame: Measured at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Referral | MBSR Referral
Number analyzed (Participants) | 12 | 6
score on a scale | 5.3 (5.4) | 3.2 (8.1)
Statistical Analysis 1: Comparison: Usual Care Referral vs MBSR Referral; Test type: Superiority; p = 0.82, t-test, 2 sided; Mean Difference (Final Values) = 3

2. Secondary Outcome: Generalized Anxiety Disorder -7
Description: Anxiety Severity by total score. Range 0-21. Mild 5-9; Moderate (10-14); Severe > 15
Time Frame: Measured at 45 days, 6 months, and 12 months
Reporting Status: Not Posted

3. Secondary Outcome: ED Utilization
Description: Return visits to the Emergency Department
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global Short Form
Description: quality of life
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Cognitive and Affective Mindfulness Scale - Revised
Description: 12-item measure (each scored 1-4) with total of 48. A higher score is consistent with greater mindfulness qualities.
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Toronto Mindfulness Scale
Description: 13-item state-mindfulness measure that has two sub-scales: Curiosity, 6 items, subscale score ranging from 0-24, and Decentering, 7 items, with a subscale score ranging from 0-28.
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Patient Health Questionnaire - 8 (Depression)
Description: Measure of current depression: None - Minimal depression (0 to 4), Mild depression (5 to 9), Moderate depression (10 to 14), Moderately severe depression (15 to 19), Severe depression (20 to 24)
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Patient Health Questionnaire - 15 (Physical Symptoms)
Description: Somatic symptom severity: Minimal 0-4, Low 5-9, Medium 10-14, High 15-30
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Healthcare Utilization
Description: Visits to care professionals other then the ED
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PTSD Screener
Description: 4 item measure (each scored 0 or 1). Higher score associated with higher likelihood of a PTSD.
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Panic Screener
Description: 5 item measure (each scored 0 or 1). Higher score associated with higher likelihood of a panic disorder.
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Social Anxiety Screener
Description: 3 item measure (each scored 1-4) with total possible score of 12. Higher score associated with higher social anxiety
Time Frame: Measured at 45 days, 3 months, 6 months, and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Usual Care Referral | MBSR Referral
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03365375/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03365375/ICF_001.pdf